CLINICAL TRIAL: NCT04587466
Title: Prospective Cohort Study of the Care Pathway for Elderly People in Care in Nursing Homes in Guadeloupe
Brief Title: KArukera Study of Aging in Nursing Homes
Acronym: KASEHPAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Agence Régionale de Santé de la Guadeloupe (Unknown)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH3_2020/04; 2020-A00960-39 (Other: ANSM)
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Geriatric Syndromes
Keywords: Older people; nursing home; hospitalization; geriatric syndromes; mortality; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nursing homes are a recent occurrence in Guadeloupe, and little is known about the characteristics of their residents. In Guadeloupe, in the French West Indies, nearly 1200 dependent older people are cared for in nursing homes. The aim of the KArukera Study of Aging in Nursing Homes (KASEHPAD) is to study the care pathways of dependent elderly people in nursing homes in Guadeloupe over a year. The main objective will be to obtain the annual rate of hospitalisation in this setting. The secondary objectives will be to assess hospitalisations costs, the incidence of mortality, the prevalence of geriatric syndromes, as well as the quality of life of residents and professional caregiver burnout. Ultimately, these results will be compared to a similar study in nursing homes, the KASAF study (for Karukera Study of Aging in Foster Families).

DETAILED DESCRIPTION:
hile not fully integrated in the Caribbean culture, nursing homes may well become a necessity, and their number is growing. For example, there are now 6 nursing homes in Jamaica, and since the first one in 1991, 20 more have opened in Guadeloupe. Being admitted in a nursing home may be beneficial for the residents as well as for their families since it offers around-the-clock medical care and a secure living environment. On the other hand, living in a nursing home also tend to alter the medical and psychological state of the resident. Little is known about the characteristics of nursing home residents in Guadeloupe. Epidemiological and medico-economic data on older people in nursing homes are essential to assess the relevance of this type of care, and several and yet unanswered questions come to mind: what is the residents' annual hospitalization rate and the associated costs? What is the prevalence of geriatric syndromes in this population, and the incidence of mortality? What is the incidence of pneumonia, the leading cause of death and emergency hospitalization in older people? What is the quality of life of the older residents and their professional caregivers? KASEHPAD, an epidemiological cohort, aims to answer these questions. This longitudinal study will assess the health status and medical and economic data of 500 nursing home residents and their professional caregivers over a year. A similar study (KASAF, for Karukera Study of Aging in Foster Families) will be conducted simultaneously among 250 older people in foster families, as to compare these two types of care.

The main outcome is the number of hospitalizations over a year. Local PMSI (Medicalization program of the information system) hospitals databases will provide information on hospital admissions.

500 people aged 60 and older and living in nursing homes in Guadeloupe will be included. Data collection will be conducted using face-to-face interviews with the participants and their professional caregivers at baseline and after 6 and 12 months, and phone interviews with the professional caregivers, after 3 and 9 months. Anthropometric measures, information on general health status and care pathways (hospitalization, medical and paramedical consultations), as well as data on medical history, cognition, nutritional status, and physical frailty will also be collected. Depressive and anxiety symptoms will also be assessed along with functional abilities (mobility, instrumental activities of daily living and activities of daily living). A systematic update of vital status (death) and care pathway will be carried out at each follow-up. Additional information on the residents' living status and potential hospitalizations will be collected after 3 and 9 months. Finally, professional caregivers will be interviewed at inclusion, after 6 months and after a year to assess their own quality of life and burnout symptoms.

This study was supported by a grant from the Agence Régionale de Santé de la Guadeloupe.

ELIGIBILITY:
Inclusion Criteria:

* participant must be over 60 years old
* residents must live in a nursing home in Guadeloupe, Saint-Martin or Saint-Barthelemy
* residents must benefit from the French social security
* Participant must have an identified support person
* Participant under guardianship or curatorship if accepted by the legal guardian
* Participant in a foreseeable short-term end-of-life situation if accepted by the legal representative or the support person

Exclusion Criteria:

* refusal from the resident or his legal guardian to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Every elderly person living in a nursing home in Guadeloupe will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-05-03 (Estimated); Study Completion 2022-11-03 (Estimated)

PRIMARY OUTCOMES:
Hospitalization rate of the participant | 12 months
  Number of hospital admissions over a year, retrieved from the local PMSI (Medicalization program of the information system) of the Hospital Center of Guadeloupe

SECONDARY OUTCOMES:
Length of hospital stays of the participant | 12 months
  Length of hospital stays expressed as number of days and nights, retrieved from the local PMSI (Medicalization program of the information system) of the Hospital Center of Guadeloupe

OTHER OUTCOMES:
Medical consultations of the participant | inclusion
  Number of consultations with a general practitioner, a medical specialist or paramedical professional will be collected.
  This information will be retrieved from the CRF using the RUD-Lite scale (Resource Utilization in Dementia questionnaire). This scale assesses the use of healthcare resources by people suffering from dementia. The professional caregiver will complete this questionnaire at inclusion.
Medical consultations of the participant | 3 months
  Number of consultations with a general practitioner, a medical specialist or paramedical professional will be collected.
  This information will be retrieved from the CRF using the RUD-Lite scale (Resource Utilization in Dementia questionnaire). This scale assesses the use of healthcare resources by people suffering from dementia. The professional caregiver will complete this questionnaire at the 3-month follow-up.
Medical consultations of the participant | 6 months
  Number of consultations with a general practitioner, a medical specialist or paramedical professional will be collected.
  This information will be retrieved from the CRF using the RUD-Lite scale (Resource Utilization in Dementia questionnaire). This scale assesses the use of healthcare resources by people suffering from dementia. The professional caregiver will complete this questionnaire at the 6-month follow-up.
Medical consultations of the participant | 9 months
  Number of consultations with a general practitioner, a medical specialist or paramedical professional will be collected.
  This information will be retrieved from the CRF using the RUD-Lite scale (Resource Utilization in Dementia questionnaire). This scale assesses the use of healthcare resources by people suffering from dementia. The professional caregiver will complete this questionnaire at the 9-month follow-up.
Medical consultations of the participant | 12 months
  Number of consultations with a general practitioner, a medical specialist or paramedical professional will be collected.
  This information will be retrieved from the CRF using the RUD-Lite scale (Resource Utilization in Dementia questionnaire). This scale assesses the use of healthcare resources by people suffering from dementia. The professional caregiver will complete this questionnaire at the 12-month follow-up.
Global cost of hospitalization of the participant | 12 months
  Global cost of hospitalization will be retrieved from the local PMSI (Medicalization program of the information system) databases after study completion
Vital status of the participant | 3 months
  Vital status (alive or deceased) will be collected at the 3-month follow-up from the professional caregiver.
Vital status of the participant | 6 months
  Vital status (alive or deceased) will be collected at the 6-month follow-up from the professional caregiver.
Vital status of the participant | 9 months
  Vital status (alive or deceased) will be collected at the 9-month follow-up , from the professional caregiver.
Vital status of the participant | 12 months
  Vital status (alive or deceased) will be collected at the 12-month follow-up , from the professional caregiver.
Lower respiratory tract infections of the participant | inclusion
  Occurrence of lower respiratory tract infections will be collected using the RUD-lite. For the diagnosis of lower respiratory tract infections, at least two of the following must be present and a doctor must confirm the clinical evidence: Cough (starting or worsening) that may produce phlegm, specific clinical signs during auscultation; Fever. (≥38°C); Chest pain ; Rapid, shallow breathing ((≥25 per minute) ; Confusion or increased dependency.
  The professional caregiver will complete this question at inclusion.
Lower respiratory tract infections of the participant | 3 months
  Occurrence of lower respiratory tract infections will be collected using the RUD-lite. For the diagnosis of lower respiratory tract infections, at least two of the following must be present and a doctor must confirm the clinical evidence: Cough (starting or worsening) that may produce phlegm, specific clinical signs during auscultation; Fever. (≥38°C); Chest pain ; Rapid, shallow breathing ((≥25 per minute) ; Confusion or increased dependency.
  The professional caregiver will complete this question at the 3-month follow-up.
Lower respiratory tract infections of the participant | 6 months
  Occurrence of lower respiratory tract infections will be collected using the RUD-lite. For the diagnosis of lower respiratory tract infections, at least two of the following must be present and a doctor must confirm the clinical evidence: Cough (starting or worsening) that may produce phlegm, specific clinical signs during auscultation; Fever. (≥38°C); Chest pain ; Rapid, shallow breathing ((≥25 per minute) ; Confusion or increased dependency.
  The professional caregiver will complete this question at the 6-month follow-up.
Lower respiratory tract infections of the participant | 9 months
  Occurrence of lower respiratory tract infections will be collected using the RUD-lite. For the diagnosis of lower respiratory tract infections, at least two of the following must be present and a doctor must confirm the clinical evidence: Cough (starting or worsening) that may produce phlegm, specific clinical signs during auscultation; Fever. (≥38°C); Chest pain ; Rapid, shallow breathing ((≥25 per minute) ; Confusion or increased dependency.
  The professional caregiver will complete this question at the 9-month follow-up.
Lower respiratory tract infections of the participant | 12 months
  Occurrence of lower respiratory tract infections will be collected using the RUD-lite. For the diagnosis of lower respiratory tract infections, at least two of the following must be present and a doctor must confirm the clinical evidence: Cough (starting or worsening) that may produce phlegm, specific clinical signs during auscultation; Fever. (≥38°C); Chest pain ; Rapid, shallow breathing ((≥25 per minute) ; Confusion or increased dependency.
  The professional caregiver will complete this question at at the 12-month follow-up.
Falls of the participant | 6 months
  Total number of falls since the last visit will be collected at the 6-month follow-up from the professional caregivers.
Falls of the participant | 12 months
  Total number of falls since the last visit will be collected at the 12-month follow-up from the professional caregivers.
Cognition of the participant | inclusion
  The level of cognitive deterioration of the participants will be with the Mini Mental State Examination (MMSE). This 30-item scale assesses the severity of cognitive deterioration through items of orientation, learning, attention and arithmetic, memory, language, and constructive praxis.
  The scale is rated from 0 to 30, reflecting the level of cognitive impairment. The participant will complete this questionnaire at inclusion.
Cognition of the participant | 6 months
  The level of cognitive deterioration of the participants will be with the Mini Mental State Examination (MMSE). This 30-item scale assesses the severity of cognitive deterioration through items of orientation, learning, attention and arithmetic, memory, language, and constructive praxis.
  The scale is rated from 0 to 30, reflecting the level of cognitive impairment. The participant will complete this questionnaire at the 6-month follow-up.
Cognition of the participant | 12 months
  The level of cognitive deterioration of the participants will be with the Mini Mental State Examination (MMSE). This 30-item scale assesses the severity of cognitive deterioration through items of orientation, learning, attention and arithmetic, memory, language, and constructive praxis.
  The scale is rated from 0 to 30, reflecting the level of cognitive impairment. The participant will complete this questionnaire at the 12-month follow-up.
Depressive symptoms of the participant | inclusion
  Depressive symptoms will be assessed using the CES-D (Center for Epidemiologic Studies- Depression Scale validated in French by Fuhrer & Rouillon This 20-item questionnaire assesses depressive symptomatology, including 4 items on positive affect (happiness, self-worth, confidence, enjoyment). Frequency of symptom occurrence during the past week is assessed by the participant using a 4-point Likert scale ("never", "occasionally", "quite often" and "frequently"). The score ranges from 0 to 60. The higher the score, the more significant the symptomatology. Data will be collected at inclusion, T6 and T12. For statistical analyses, the variable will be dichotomized (1 = presence of depression and 0 = absence of depression). The participant will complete this questionnaire at inclusion.
Depressive symptoms of the participant | 6 months
  Depressive symptoms will be assessed using the CES-D (Center for Epidemiologic Studies- Depression Scale validated in French by Fuhrer & Rouillon This 20-item questionnaire assesses depressive symptomatology, including 4 items on positive affect (happiness, self-worth, confidence, enjoyment). Frequency of symptom occurrence during the past week is assessed by the participant using a 4-point Likert scale ("never", "occasionally", "quite often" and "frequently"). The score ranges from 0 to 60. The higher the score, the more significant the symptomatology. Data will be collected at inclusion, T6 and T12. For statistical analyses, the variable will be dichotomized (1 = presence of depression and 0 = absence of depression). The participant will complete this questionnaire at the 6-month follow-up
Depressive symptoms of the participant | 12 months
  Depressive symptoms will be assessed using the CES-D (Center for Epidemiologic Studies- Depression Scale validated in French by Fuhrer & Rouillon This 20-item questionnaire assesses depressive symptomatology, including 4 items on positive affect (happiness, self-worth, confidence, enjoyment). Frequency of symptom occurrence during the past week is assessed by the participant using a 4-point Likert scale ("never", "occasionally", "quite often" and "frequently"). The score ranges from 0 to 60. The higher the score, the more significant the symptomatology. Data will be collected at inclusion, T6 and T12. For statistical analyses, the variable will be dichotomized (1 = presence of depression and 0 = absence of depression). The participant will complete this questionnaire at the 12-month follow-up.
Feeling of loneliness of the participant | inclusion
  Feeling of loneliness will be captured with the 14th item of the CES-D (14, 15): " I felt lonely ". The participant will complete this test at inclusion.
Feeling of loneliness of the participant | 6 months
  Feeling of loneliness will be captured with the 14th item of the CES-D (14, 15): " I felt lonely ". The participant will complete this test at the 6-month follow-up.
Feeling of loneliness of the participant | 12 months
  Feeling of loneliness will be captured with the 14th item of the CES-D (14, 15): " I felt lonely ". The participant will complete this test at the 12-month follow-up.
Polypharmacy of the participant | inclusion
  Total number of medications taken by participants will be collected from the professional caregiver at inclusion to assess polypharmacy.
Polypharmacy of the participant | 6 months
  Total number of medications taken by participants will be collected from the professional caregiver at the 6-month follow-up to assess polypharmacy.
Polypharmacy of the participant | 12 months
  Total number of medications taken by participants will be collected from the professional caregiver at the 12-month follow-up to assess polypharmacy.
Malnutrition of the participant | inclusion
  Malnutrition will be assessed with the short version of the Mini Nutritional Assessment (18). This questionnaire assesses nutritional status. A score under 12 indicates probable undernutrition. For the analyses, the variable will be dichotomized accordingly (1 = undernutrition; 0 = no undernutrition). The participant will complete this questionnaire at inclusion.
Malnutrition of the participant | 6 months
  Malnutrition will be assessed with the short version of the Mini Nutritional Assessment (18). This questionnaire assesses nutritional status. A score under 12 indicates probable undernutrition. For the analyses, the variable will be dichotomized accordingly (1 = undernutrition; 0 = no undernutrition). The participant will complete this questionnaire at the 6-month follow-up.
Malnutrition of the participant | 12 months
  Malnutrition will be assessed with the short version of the Mini Nutritional Assessment (18). This questionnaire assesses nutritional status. A score under 12 indicates probable undernutrition. For the analyses, the variable will be dichotomized accordingly (1 = undernutrition; 0 = no undernutrition). The participant will complete this questionnaire at the 12-month follow-up.
Sarcopenia of the participant | inclusion
  The Short Physical Performance Battery (SPPB) will help to identify sarcopenia. Three subtests measure lower-extremity functions: keeping balance (feet side-by-side, semi-tandem, tandem balance position, to be kept for 10 seconds each), walking 4 meters at usual pace, yielding a gait speed ratio (meter per second) ; standing up and sitting down five times as quickly as possible with the arms folded. Each movement is scored 0-4 points out of a total score from 0 to 12, with higher scores showing better physical performance. If total score is under 8, there is a risk of sarcopenia. For the analyses, the variable will be dichotomized accordingly (1 = sarcopenia; 0 = no sarcopenia). The participant will complete this test at inclusion.
Sarcopenia of the participant | 6 months
  The Short Physical Performance Battery (SPPB) will help to identify sarcopenia. Three subtests measure lower-extremity functions: keeping balance (feet side-by-side, semi-tandem, tandem balance position, to be kept for 10 seconds each), walking 4 meters at usual pace, yielding a gait speed ratio (meter per second) ; standing up and sitting down five times as quickly as possible with the arms folded. Each movement is scored 0-4 points out of a total score from 0 to 12, with higher scores showing better physical performance. If total score is under 8, there is a risk of sarcopenia. For the analyses, the variable will be dichotomized accordingly (1 = sarcopenia; 0 = no sarcopenia). The participant will complete this test at the 6-month follow-up.
Sarcopenia of the participant | 12 months
  The Short Physical Performance Battery (SPPB) will help to identify sarcopenia. Three subtests measure lower-extremity functions: keeping balance (feet side-by-side, semi-tandem, tandem balance position, to be kept for 10 seconds each), walking 4 meters at usual pace, yielding a gait speed ratio (meter per second) ; standing up and sitting down five times as quickly as possible with the arms folded. Each movement is scored 0-4 points out of a total score from 0 to 12, with higher scores showing better physical performance. If total score is under 8, there is a risk of sarcopenia. For the analyses, the variable will be dichotomized accordingly (1 = sarcopenia; 0 = no sarcopenia). The participant will complete this test at the 12-month follow-up.
Frailty of the participant | inclusion
  Frailty will be assessed at inclusion, T6 and T12 using Fried's phenotype (weight loss, exhaustion, low physical activity, slowness, weakness) and will be analyzed as a dichotomous variable, i.e. 1 = Fragile and 0 = Not Fragile. Information on the different components of the phenotype will be retrieved from the MNA, the SPPB and a hand-grip strength test using a dynamometer, at inclusion.
Frailty of the participant | 6 months
  Frailty will be assessed at inclusion, T6 and T12 using Fried's phenotype (weight loss, exhaustion, low physical activity, slowness, weakness) and will be analyzed as a dichotomous variable, i.e. 1 = Fragile and 0 = Not Fragile. Information on the different components of the phenotype will be retrieved from the MNA, the SPPB and a hand-grip strength test using a dynamometer, at the 6-month follow-up.
Frailty of the participant | 12 months
  Frailty will be assessed at inclusion, T6 and T12 using Fried's phenotype (weight loss, exhaustion, low physical activity, slowness, weakness) and will be analyzed as a dichotomous variable, i.e. 1 = Fragile and 0 = Not Fragile. Information on the different components of the phenotype will be retrieved from the MNA, the SPPB and a hand-grip strength test using a dynamometer, at the 12-month follow-up.
Sensory impairment of the participant | inclusion
  Sensory impairments (audition and vision) will be addressed by directly asking the professional caregiver. Variables will be dichotomized accordingly ((1 = hearing / vision impairment; 0 = hearing / vision impairment). The professional caregiver will complete this questionnaire at inclusion.
Sensory impairment of the participant | 6 months
  Sensory impairments (audition and vision) will be addressed by directly asking the professional caregiver. Variables will be dichotomized accordingly ((1 = hearing / vision impairment; 0 = hearing / vision impairment). The professional caregiver will complete this questionnaire at the 6-month follow-up.
Sensory impairment of the participant | 12 months
  Sensory impairments (audition and vision) will be addressed by directly asking the professional caregiver. Variables will be dichotomized accordingly ((1 = hearing / vision impairment; 0 = hearing / vision impairment). TThe professional caregiver will complete this questionnaire at the 12-month follow-up.
Activities of Daily Living of the participant | inclusion
  The level of independence in Activities of Daily Living (ADL) and incontinence will be assessed using the Katz's scale, a 6-item scale assessing independence in 6 basic activities of daily living: bathing, toileting, eating, dressing, incontinence. For each activity, a score of 1 indicates complete autonomy, a score of 0.5 indicates partial autonomy, and a score of 0 indicates complete dependency. The professional caregiver will complete this questionnaire about the participant at inclusion.
Activities of Daily Living of the participant | 6 months
  The level of independence in Activities of Daily Living (ADL) and incontinence will be assessed using the Katz's scale, a 6-item scale assessing independence in 6 basic activities of daily living: bathing, toileting, eating, dressing, incontinence. For each activity, a score of 1 indicates complete autonomy, a score of 0.5 indicates partial autonomy, and a score of 0 indicates complete dependency. The professional caregiver will complete this questionnaire about the participant at the 6-month follow-up.
Activities of Daily Living of the participant | 12 months
  The level of independence in Activities of Daily Living (ADL) and incontinence will be assessed using the Katz's scale, a 6-item scale assessing independence in 6 basic activities of daily living: bathing, toileting, eating, dressing, incontinence. For each activity, a score of 1 indicates complete autonomy, a score of 0.5 indicates partial autonomy, and a score of 0 indicates complete dependency. The professional caregiver will complete this questionnaire about the participant at the 12-month follow-up.
Instrumental Activities of Daily Living of the participant | inclusion
  The level of independence in Instrumental Activities of Daily Living (IADL) will be assessed using Lawton's IADL scale. The professional caregiver will complete this questionnaire about the participant at inclusion.
Instrumental Activities of Daily Living of the participant | 6 months
  The level of independence in Instrumental Activities of Daily Living (IADL) will be assessed using Lawton's IADL scale. The professional caregiver will complete this questionnaire about the participant at the 6-month follow-up.
Instrumental Activities of Daily Living of the participant | 12 months
  The level of independence in Instrumental Activities of Daily Living (IADL) will be assessed using Lawton's IADL scale. The professional caregiver will complete this questionnaire about the participant at the 12-month follow-up.
Dependency of the participant | inclusion
  In France, the AGGIR questionnaire has been developed by public authorities to quickly assess the degree of dependency of elderly people, and assign a dependency group, ranging from 0 (bedridden, completely dependent) to 6 (no help required, the person is autonomous in everyday activities.) This scale is routinely completed by every nursing home at admission and updated when necessary to reassess healthcare pathways. The professional caregiver will complete this questionnaire about the participant at inclusion.
Dependency of the participant | 6 months
  In France, the AGGIR questionnaire has been developed by public authorities to quickly assess the degree of dependency of elderly people, and assign a dependency group, ranging from 0 (bedridden, completely dependent) to 6 (no help required, the person is autonomous in everyday activities.) This scale is routinely completed by every nursing home at admission and updated when necessary to reassess healthcare pathways. The professional caregiver will complete this questionnaire about the participant at the 6-month follow-up.
Dependency of the participant | 12 months
  In France, the AGGIR questionnaire has been developed by public authorities to quickly assess the degree of dependency of elderly people, and assign a dependency group, ranging from 0 (bedridden, completely dependent) to 6 (no help required, the person is autonomous in everyday activities.) This scale is routinely completed by every nursing home at admission and updated when necessary to reassess healthcare pathways. The professional caregiver will complete this questionnaire about the participant at at the 12-month follow-up.
Psychological and Behavioral Symptoms in Dementia of the participant | inclusion
  Psychological and Behavioral Symptoms in Dementia will be assessed with the short version of the NeuroPsychiatric Inventory or NPI. This scale assesses presence, severity for the patient and impact on the professional's workload of an array of psychological and behavioral manifestations (agitation, hallucinations, apathy, etc.) as well as neurovegetative symptoms (sleep and appetite). The professional caregiver will complete this questionnaire about the participant at inclusion.
Psychological and Behavioral Symptoms in Dementia of the participant | 6 months
  Psychological and Behavioral Symptoms in Dementia will be assessed with the short version of the NeuroPsychiatric Inventory or NPI. This scale assesses presence, severity for the patient and impact on the professional's workload of an array of psychological and behavioral manifestations (agitation, hallucinations, apathy, etc.) as well as neurovegetative symptoms (sleep and appetite). The professional caregiver will complete this questionnaire about the participant at the 6-month follow-up.
Psychological and Behavioral Symptoms in Dementia of the participant | 12 months
  Psychological and Behavioral Symptoms in Dementia will be assessed with the short version of the NeuroPsychiatric Inventory or NPI. This scale assesses presence, severity for the patient and impact on the professional's workload of an array of psychological and behavioral manifestations (agitation, hallucinations, apathy, etc.) as well as neurovegetative symptoms (sleep and appetite). The professional caregiver will complete this questionnaire about the participant at the 12-month follow-up.
Risk of developing pressure ulcers of the participant | inclusion
  Risk of developing pressure ulcers will be assessed with the Braden's Scale, and pressure ulcers will be classified according to the National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance. The professional caregiver will complete this questionnaire about the participant at inclusion.
Risk of developing pressure ulcers of the participant | 6 months
  Risk of developing pressure ulcers will be assessed with the Braden's Scale, and pressure ulcers will be classified according to the National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance. The professional caregiver will complete this questionnaire about the participant at the 6-month follow-up.
Risk of developing pressure ulcers of the participant | 12 months
  Risk of developing pressure ulcers will be assessed with the Braden's Scale, and pressure ulcers will be classified according to the National Pressure Ulcer Advisory Panel, European Pressure Ulcer Advisory Panel and Pan Pacific Pressure Injury Alliance. The professional caregiver will complete this questionnaire about the participant at the 12-month follow-up.
Quality of life of the participant | inclusion
  Quality of life of the participant will be assessed using the QoL-AD (Questionnaire Quality of Life - Alzheimer's Disease). This 13-item questionnaire assesses the participant's physical condition, mood, relationships with friends and family, financial difficulties, and overall quality of life. The self-rated and the proxy-rated version of the questionnaire will be administered to the participant and the caregiver, respectively. The items are evaluated using a 4-point ordinal scale ranging from poor to excellent, with a total score ranging from 13 to 52. For the weighted score, the participant's score is multiplied by 2, the caregiver's score (about the participant's quality of life) is added, and the total is divided by 3 to bring the score back to the initial scale. The participant and the professional caregiver will complete this test at inclusion.
Quality of life of the participant | 6 months
  Quality of life of the participant will be assessed using the QoL-AD (Questionnaire Quality of Life - Alzheimer's Disease). This 13-item questionnaire assesses the participant's physical condition, mood, relationships with friends and family, financial difficulties, and overall quality of life. The self-rated and the proxy-rated version of the questionnaire will be administered to the participant and the caregiver, respectively. The items are evaluated using a 4-point ordinal scale ranging from poor to excellent, with a total score ranging from 13 to 52. For the weighted score, the participant's score is multiplied by 2, the caregiver's score (about the participant's quality of life) is added, and the total is divided by 3 to bring the score back to the initial scale. The participant and the professional caregiver will complete this test at the 6-month follow-up.
Quality of life of the participant | 12 months
  Quality of life of the participant will be assessed using the QoL-AD (Questionnaire Quality of Life - Alzheimer's Disease). This 13-item questionnaire assesses the participant's physical condition, mood, relationships with friends and family, financial difficulties, and overall quality of life. The self-rated and the proxy-rated version of the questionnaire will be administered to the participant and the caregiver, respectively. The items are evaluated using a 4-point ordinal scale ranging from poor to excellent, with a total score ranging from 13 to 52. For the weighted score, the participant's score is multiplied by 2, the caregiver's score (about the participant's quality of life) is added, and the total is divided by 3 to bring the score back to the initial scale. The participant and the professional caregiver will complete this test at the 12-month follow-up.
Health-related quality of life of the participant | inclusion
  Health-related quality of life of the participant will be assessed with the EQ-5D questionnaire. This questionnaire assesses health conditions. It is the most widely used questionnaire in medico-economic analyses. It allows health outcomes to be assessed in terms of QALYs (Quality-Adjusted Life-Years). This indicator summarizes the length and quality of life in a single figure. The result of a cost-utility analysis is expressed in terms of the cost of gaining one QALY (i.e. one year lived in perfect health). To estimate QALY, health-related quality of life is designed on a continuum from 0 (death) to 1 (perfect health). Each health status is thus assigned a weight of 0 to 1, the higher the corresponding quality of life.
  The participant and the foster caregiver will complete this test at inclusion.
Health-related quality of life of the participant | 6 months
  Health-related quality of life of the participant will be assessed with the EQ-5D questionnaire. This questionnaire assesses health conditions. It is the most widely used questionnaire in medico-economic analyses. It allows health outcomes to be assessed in terms of QALYs (Quality-Adjusted Life-Years). This indicator summarizes the length and quality of life in a single figure. The result of a cost-utility analysis is expressed in terms of the cost of gaining one QALY (i.e. one year lived in perfect health). To estimate QALY, health-related quality of life is designed on a continuum from 0 (death) to 1 (perfect health). Each health status is thus assigned a weight of 0 to 1, the higher the corresponding quality of life.
  The participant and the foster caregiver will complete this test at the 6-month follow-up.
Health-related quality of life of the participant | 12 months
  Health-related quality of life of the participant will be assessed with the EQ-5D questionnaire. This questionnaire assesses health conditions. It is the most widely used questionnaire in medico-economic analyses. It allows health outcomes to be assessed in terms of QALYs (Quality-Adjusted Life-Years). This indicator summarizes the length and quality of life in a single figure. The result of a cost-utility analysis is expressed in terms of the cost of gaining one QALY (i.e. one year lived in perfect health). To estimate QALY, health-related quality of life is designed on a continuum from 0 (death) to 1 (perfect health). Each health status is thus assigned a weight of 0 to 1, the higher the corresponding quality of life.
  The participant and the foster caregiver will complete this test at the 12-month follow-up.
Adaptation to the nursing home of the participant | inclusion
  Adaptation to the professional family will be assessed using Castonguay & Ferron's scale. This is a 17-item scale designed to identify people who have difficulties to adjust to nursing home life. The participants must answer "yes" or "no" to a series of statements about their daily life and habits in the residence. A score of 16 or 17 indicates a good general adaptation, while a score of 11 or less indicates significant difficulties. The participant and the professional caregiver will complete this test at inclusion.
Adaptation to the nursing home of the participant | 6 months
  Adaptation to the professional family will be assessed using Castonguay & Ferron's scale. This is a 17-item scale designed to identify people who have difficulties to adjust to nursing home life. The participants must answer "yes" or "no" to a series of statements about their daily life and habits in the residence. A score of 16 or 17 indicates a good general adaptation, while a score of 11 or less indicates significant difficulties. The participant and the professional caregiver will complete this test at the 6-month follow-up.
Adaptation to the nursing home of the participant | 12 months
  Adaptation to the professional family will be assessed using Castonguay & Ferron's scale. This is a 17-item scale designed to identify people who have difficulties to adjust to nursing home life. The participants must answer "yes" or "no" to a series of statements about their daily life and habits in the residence. A score of 16 or 17 indicates a good general adaptation, while a score of 11 or less indicates significant difficulties. The participant and the professional caregiver will complete this test at the 12-month follow-up.
Professional caregivers' quality of life assessed with SF-36 | inclusion
  Professional caregivers' quality of life will be assessed with the Medical Outcomes Study Short-Form General Health Survey - 36 items (SF-36, a widely validated health-related quality of life questionnaire, that uses questions on physical, social and psychological domains. The professional caregiver will complete this questionnaire at inclusion.
Professional caregivers' quality of life assessed with SF-36 | 6 months
  Professional caregivers' quality of life will be assessed with the Medical Outcomes Study Short-Form General Health Survey - 36 items (SF-36, a widely validated health-related quality of life questionnaire, that uses questions on physical, social and psychological domains. The professional caregiver will complete this questionnaire at the 6-month follow-up.
Professional caregivers' quality of life assessed with SF-36 | 12 months
  Professional caregivers' quality of life will be assessed with the Medical Outcomes Study Short-Form General Health Survey - 36 items (SF-36, a widely validated health-related quality of life questionnaire, that uses questions on physical, social and psychological domains. The professional caregiver will complete this questionnaire at the 12-month follow-up.
Professional caregivers' quality of life assessed with the Pro-QoL scale | inclusion
  Symptoms of burnout will be assessed with the Pro-QoL scale (professional quality of life scale). This 30-item questionnaire yields three domain-specific scores: burnout risk, compassion, and compassion fatigue. The professional caregiver will complete this questionnaire at inclusion.
Professional caregivers' quality of life assessed with the Pro-QoL scale | 6 months
  Symptoms of burnout will be assessed with the Pro-QoL scale (professional quality of life scale). This 30-item questionnaire yields three domain-specific scores: burnout risk, compassion, and compassion fatigue. The professional caregiver will complete this questionnaire at the 6-month follow-up.
Professional caregivers' quality of life assessed with the Pro-QoL scale | 12 months
  Symptoms of burnout will be assessed with the Pro-QoL scale (professional quality of life scale). This 30-item questionnaire yields three domain-specific scores: burnout risk, compassion, and compassion fatigue. The professional caregiver will complete this questionnaire at the 12-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Maturin MT TABUE-TEGUO, MD MhD, Principal Investigator — CHU de la Guadeloupe
Locations (11):
- Guadeloupe (10):
  - Ehpad Residence Sacré Cœur, Basse-Terre
  - Ehpad Nou Gran Moun, Capesterre-Belle-Eau
  - Ehpad Residence Senior 'Les Flamboyants', Gourbeyre
  - Ehpad St-Christophe, Grand-Bourg
  - Ehpad Domaine de Choisy, Le Gosier
  - Ehpad Ch Jacques Salin, Les Abymes
  - Ehpad Les Jardins de Belost, Saint-Claude
  - Ehpad Res. Medico-Sle de Marie-Galante, Saint-Louis
  - Ehpad Les Roses de Lima, Sainte-Rose
  - Ehpad Kalana, Village
- Ehpad Bethany Home, Saint Martin, Saint Martin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boucaud-Maitre D, Amieva H, Pic O, Letchimy L, Simo N, Dartigues JF, Drame M, Dorey JM, Tabue-Teguo M. Poor adjustment to nursing homes and 1-year mortality: a secondary analysis of the KASEHPAD cohort study. BMJ Open. 2025 Dec 4;15(12):e106682. doi: 10.1136/bmjopen-2025-106682. PMID 41344708